CLINICAL TRIAL: NCT04649541
Title: An Adaptive, Randomized, Double Blind, Placebo Controlled Three Part Study of the Safety, Tolerability, and Pharmacokinetics of MRX-8 Administered Intravenously to Healthy Volunteers in Single Ascending and Multiple Ascending Dose Cohorts
Brief Title: Study of the Safety, Tolerability, and PK of MRX-8 Administered Intravenously to HVs in SAD and MAD Cohorts
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MicuRx (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRX8-101
Record Dates: First submitted 2020-11-16; First posted 2020-12-02 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Single intravenous doses of MRX-8 (Active Comparator): Single escalating doses of MRX-8
  Interventions: Drug: MRX-8
- Single intravenous doses of placebo (Placebo Comparator): Single intravenous doses of placebo to match MRX-8
  Interventions: Drug: Placebo
- Multiple intravenous doses of MRX-8 for 7 days (Active Comparator): Multiple ascending intravenous doses of MRX-8 every 12 hours for 7 days.
  Interventions: Drug: MRX-8
- Multiple intravenous doses of placebo for 7 days (Placebo Comparator): Multiple intravenous doses of placebo every 12 hours for 7 days to match MRX-8.
  Interventions: Drug: Placebo
- Multiple intravenous doses of MRX-8 for 14 days (Active Comparator): Multiple ascending intravenous doses of MRX-8 every 12 hours for 14 days.
  Interventions: Drug: MRX-8
- Multiple intravenous doses of placebo for 14 days (Placebo Comparator): Multiple intravenous doses of placebo every 12 hours for 14 days to match MRX-8.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MRX-8 — novel semi-synthetic polymyxin B analog.
  Arms: Multiple intravenous doses of MRX-8 for 14 days; Multiple intravenous doses of MRX-8 for 7 days; Single intravenous doses of MRX-8
Drug: Placebo — 5% dextrose in water
  Arms: Multiple intravenous doses of placebo for 14 days; Multiple intravenous doses of placebo for 7 days; Single intravenous doses of placebo

SUMMARY:
This Phase 1 study is designed to assess the safety and tolerability of single and multiple intravenous (IV) doses of MRX-8, to assess the pharmacokinetics of MRX-8 and its primary metabolite following single and multiple IV doses, and to measure the elimination of MRX-8 and its metabolite in urine.

DETAILED DESCRIPTION:
This is a first-in-human, randomized, double-blind, placebo-controlled study consisting of 3 parts. Part 1 will evaluate single ascending doses (SAD) of study drug. Part 2 will evaluate multiple ascending doses (MAD) of study drug administered for 7 days. Part 3 will evaluate MAD of study drug administered for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* In good general health

Exclusion Criteria:

* Prior participation in a study utilizing a polymyxin or aminoglycoside antibiotic or other nephrotoxic drug within the 12 months prior to study drug administration on Day 1
* Use of tobacco or nicotine products, in any form, within 30 days prior to study drug administration on Day 1
* Venous access considered inadequate for IV infusions, laboratory safety assessments, or PK sample collection
* Underlying hepatic, renal, metabolic, cardiovascular or immunologic disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2020-11-29 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | Pre-dose through 48 hours after the end of infusion on the final infusion of study drug
  Symptoms reported by subjects.
Clinical laboratory assessment | Pre-dose through 48 hours after the end of infusion on the final infusion of study drug
  Complete blood count
Peak Plasma Concentration (Cmax) | Pre-dose through 48 hours after the end of infusion on the final infusion of study drug
  Cmax of MRX-8 and its primary metabolite following single and multiple intravenous doses
Time to Peak Plasma Concentration (Tmax) | Pre-dose through 48 hours after the end of infusion on the final infusion of study drug
  Tmax of MRX-8 and its primary metabolite following single and multiple intravenous doses
Area under the plasma concentration versus time curve (AUC) | Pre-dose through 48 hours after the end of infusion on the final infusion of study drug
  AUC of MRX-8 and its primary metabolite following single and multiple intravenous doses
Vital signs | Pre-dose through 48 hours after the end of infusion on the final infusion of study drug
  Heart rate

SECONDARY OUTCOMES:
Elimination of MRX-8 and its primary metabolite in urine | At the end of infusion through 24 hours after the end of infusion on the final infusion of study drug
  Quantity of measurable MRX-8 and its primary metabolite excreted in urine

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No